CLINICAL TRIAL: NCT04449146
Title: Scapular Positioning in Standing Position Using Sonography
Acronym: 3S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3S (29BRC18.0239)
Record Dates: First submitted 2019-10-29; First posted 2020-06-26 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Shoulder Osteoarthritis; Arthropathy Shoulder
Keywords: Reverse Shoulder Arthroplasty

STUDY DESIGN:
Intervention Model Description: This is mono-center study. Patients in the process of preoperative care of a Reverse Shoulder Arthroplasty (CT Scan already available as part of the extended care course) will be offered the study. A localizer ultrasound will be performed during surgical consultation or the day before the surgical procedure in standing position (duration: 1/2 day).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- shoulder localizer ultrasound (Experimental): The localizer ultrasound of the shoulder is performed on an unclothed patient (at the shoulders) and comes to locate bony landmarks using the ultrasound probe as a Transcutaneous localizer. The Protocol plans to acquire different landmarks on the scapula: lower angle, coracoid, scapula spine and bilateral acromioclavicular joint (definition of the coronal plan). These acquisitions are carried out by the probe connected to a Tablet (Microsoft surface Pro 3) which allows to locate the probe and by extension of the probe the location of the points selected by ultrasound.
  Interventions: Diagnostic Test: Scapular positioning in Standing position using Sonography

INTERVENTIONS:
Diagnostic Test: Scapular positioning in Standing position using Sonography — The localizer ultrasound of the shoulder is performed in an unclothed patient (at the shoulders) and comes to locate bony landmarks using the ultrasound probe as a Transcutaneous localizer.

SUMMARY:
The objective of this study is to analyse the positioning of the scapula in standing position and compared to the supine position (CT scan) in 3 dimensions (3 rotations of the scapula) using a non-radiant, portable system, combining an ultrasound probe with marker and a camera integrated into a Tablet for the three-dimensional location of the marker (probe).

DETAILED DESCRIPTION:
This is a mono-center trial. Patients in the process of pre-operative care of a reverse shoulder arthroplasty (CT Scan already available as part of the care course in supine position) will be offered the study. A localizer ultrasound will be performed during surgical consultation or the day before the surgery in standing position (duration: 1/2 day). This consultation takes place during the course of the surgical consultation or when the patient is admitted the day before his surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Major patients and agreeing to participate in the study after oral and written information.
* Care course patients for a reverse shoulder arthroplasty on a native shoulder joint

Exclusion Criteria:

* Patients under the age of 18
* Patients refusing to participate in the study
* Patients whose condition does not allow informed consent
* Patients who are subject to legal protection (safeguarding of Justice, curatorship, guardianship), persons deprived of their liberty
* Unaffiliated patients and non-beneficiaries of a health insurance plan

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Study the location of the scapula in 3 dimensions for the patient in standing position | Day 1
  descriptive statistics of the population : mean and standard deviation of the 3 rotations of the scapula in each plane of reference coronal plane expressed in degree.
  Comparison with the supine position and analysis of any differences.
Study the location of the scapula in 3 dimensions for the patient in standing position | Day1
  descriptive statistics of the population : mean and standard deviation of the 3 rotations of the scapula in each plane of reference axial plane expressed in degree.
  Comparison with the supine position and analysis of any differences.
Study the location of the scapula in 3 dimensions for the patient in standing position | Day 1
  descriptive statistics of the population : mean and standard deviation of the 3 rotations of the scapula in each plane of reference sagittal plane expressed in degree.
  Comparison with the supine position and analysis of any differences.

SECONDARY OUTCOMES:
Evaluating the accuracy of the device using a validation bench | Day 1
  Validation of the device using a biomechanical bench. The rotation will be assessed in coronal plane in degree. The differences between the measurements of the biomechanical bench will be compared to the measurements validation bench to assess the mean error and standard deviation of the ultrasound device
Evaluating the accuracy of the device using a validation bench | Day 1
  Validation of the device using a biomechanical bench. The rotation will be assessed in axial plane in degree. The differences between the measurements of the biomechanical bench will be compared to the measurements validation bench to assess the mean error and standard deviation of the ultrasound device
Evaluating the accuracy of the device using a validation bench | Day 1
  Validation of the device using a biomechanical bench. The rotation will be assessed in sagittal plane in degree. The differences between the measurements of the biomechanical bench will be compared to the measurements validation bench to assess the mean error and standard deviation of the ultrasound device

CONTACTS AND LOCATIONS:
Overall Officials: Hoel LETISSIER, Dr, Principal Investigator — University Hospital, Brest
Locations (1):
- Brest, University Hospital, Brest, France

IPD SHARING:
Plan to Share IPD: No